CLINICAL TRIAL: NCT01893749
Title: Primary Care Internet Based Depression Prevention for Adolescents (Promoting AdolescenT Health-PATH)
Brief Title: Primary Care Internet Based Depression Prevention for Adolescents (CATCH-IT) Also Known as Promoting AdolescenT Health
Acronym: CATCH-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin Van Voorhees, MD, MPH (Other)
Collaborators: Wellesley College (Other); Northwestern University (Other); Harvard Vanguard Medical Associates (Other); Access Healthcare Systems (Other); Endeavor Health (Other); Infant Welfare Society (Unknown); Wake Forest University Health Sciences (Other); Franciscan St. Margaret Health - Franciscan Alliance (Unknown)
Responsible Party: Sponsor-Investigator, Benjamin Van Voorhees, MD, MPH, Associate Professor of Medicine, Chief, Section of General Pediatrics and Adolescent Medicine, TIKES Center Director, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011-0505; 1R01MH090035-01A1 (NIH)
Record Dates: First submitted 2012-06-05; First posted 2013-07-09 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Major Depression; Depressive Episodes
Keywords: depression; prevention; teen; at risk; internet
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CATCH-IT (Experimental): 200 randomized teens 13-18 year old (inclusive) will be enrolled into the online program that contains 14 modules focused various therapeutic techniques, a booster session of 6 modules at the end of the online program and three 15 minute visits with their primary care doctor to discuss the benefits and disadvantages of the program.
  Parents will also be invited to participant in a partnering online program involving 4 modules online and 1 optional module. They will be asked to then participate in three 15 minute interviews with a member of the study team to discuss the benefits and disadvantages of the program.
  Interventions: Behavioral: CATCH-IT
- Health Education (No Intervention): 200 randomized teens, ages 13-18 year old (inclusive) receiving an online program with 14 modules that focus on general health education, depression, diet, exercise, hygiene and safety.
  Parents will also be invited to participate in an online program with 4 modules that also focus on general health education.

INTERVENTIONS:
Behavioral: CATCH-IT — It contains 14 modules focused on behavioral activation, cognitive behavioral therapy, interpersonal therapy and a resiliency building model, including elements such as narratives, video diaries, skill building exercises and a booster program (not yet initiated) with 6 modules that involves interaction with a live therapist. It also includes three 15-minute meetings with the primary care provider at baseline, 2 months and 12 months post intervention. These meetings are focused on the motivational interview approach where the patient and the doctor talk about the mental/physical health goals of the patient and determine the best approach for the patient by allowing the patient to have full input into the plan.
  Other Names: CATCH-IT 2; CATCH-IT 3
  Arms: CATCH-IT

SUMMARY:
The purpose of this randomized multiple-site clinical study is to determine whether a revised CATCH-IT (Internet-based depression prevention program) is more effective than a general health education Internet intervention (Health Education)on teens ages 13-18 (inclusive). It is hypothesized that teens in CATCH-IT will exhibit lower levels of depressed mood and/or maintain lower depressive scores over 2 years long-term follow up as compared to teens in Health Education group.

DETAILED DESCRIPTION:
Additional aims and hypothesis are provided below:

-Aim 1: To determine whether the CATCH-IT depression prevention intervention prevents or delays major depressive episodes, as well as non-affective disorder episodes, compared to HEALTH EDUCATION.

Hypothesis 1: Compared to youth in the HEALTH EDUCATION condition, youth assigned to CATCH-IT will have a lower hazard ratio of major depressive episodes and non-affective disorder episodes over 2 years.

-Aim 2: To determine if participants in the CATCH-IT group exhibit more rapid favorable changes of depressive symptoms/and or vulnerability/protective factors compared to the HEALTH EDUCATION group.

Hypothesis 2: Compared to youth in the HEALTH EDUCATION condition, youth in the CATCH-IT program will demonstrate a steeper slope of improved symptoms and fewer depressed days over 2 years.

-Aim 3: To determine if participants in the CATCH-IT program report lower perceived educational impairment, greater quality of life, greater health-related quality of life, and lower incidence of other mental disorders (anxiety, substance/alcohol use) as compared to participants in HEALTH EDUCATION.

Hypothesis 3: Compared to youth in the HEALTH EDUCATION group, youth in the CATCH-IT program will demonstrate more rapid benefits in reduced educational impairment, improved quality of life, and fewer disorders over 2 years.

-Aim 4: To determine for whom (moderators)among 13-18 year old (inclusive) and how (mediators) the CATCH-IT program works.

Hypothesis 4.1: CATCH-IT effects will be moderated by six domains: (1) demographic/cultural factors, (2) vulnerability factors/adverse events,(3) motivation,(4) physician relationship, (5) parent/child co-morbid psychopathology, and (6) treatment.

Hypothesis 4.2: The relation between CATCH-IT participation and reduction in depressive episodes will be mediated by adherence to the Internet, motivational interview fidelity as they alter vulnerability factors (e.g. motivation, cognition and social support) and responses to adverse events, which in turn impact the likelihood of episodes.

Exploratory Aim 1: To determine the implementation feasibility of the intervention from the physician/nurse practitioner and office nurse/medical assistant perspective as well as to describe the practices in relationship to the medical home model.

Exploratory Aim 2: To determine whether CATCH-IT has a favorable cost-benefit ratio and/or cost effectiveness of <$50,000/disability adjusted life year compared to the HEALTH EDUCATION group.

ELIGIBILITY:
Inclusion Criteria:

Adolescents:

(A) Youth ages 13 through 18 who are English speaking. (B) Youth must be experiencing elevated level of depressive symptoms on the Center for Epidemiologic Studies Depression (CES-D) scale (score >/= 16). (C) Youth will be included if they have a past history of depression, anxiety, externalizing symptoms, or substance abuse. Youth presenting in partial remission from a major depressive episode at Baseline will be rescreened after 2 months utilizing the phone screen to ensure episode is fully remitted prior to randomization or access to study intervention. Those who do not fully remit after two months will be excluded.

Parents:

*Parent of eligible adolescents

Physicians (PCP) or NP:

*Physician in any of the study sites

Healthcare Professionals:

*Primary care practice for a minimum of 6 months

Exclusion Criteria:

Adolescents:

* Current DSM-IV diagnosis of Major Depressive Disorder
* Current therapy for depression, or be taking antidepressants (e.g., SSRIs, TCAs, MAOIs, bupropion, nefazodone, mirtazapine, venlafaxine);
* Current CES-D score >35;
* DSM-IV diagnosis of schizophrenia (current or past) or bipolar affective disorder;
* Current serious medical illness that causes significant disability or dysfunction;
* Significant reading impairment (a minimum sixth-grade reading level based on parental report), mental retardation, or developmental disabilities;
* Serious imminent suicidal risk (as determined by endorsement of current suicide on CES-D or in KSADS interview) or other conditions that may require immediate psychiatric hospitalization
* Psychotic features or disorders, or currently be receiving psychotropic medication
* Extreme, current drug/alcohol abuse (greater than or equal to 2 on the CRAFFT).

Parents:

* Ineligible child
* Non-English speaking

Physicians:

*None

Healthcare Professionals:

*None

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1142 (Actual)
Dates: Start 2012-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Major Depressive Episode (major and sub-threshold) | 0, 2, 6, 12, 18 and 24 months
  Kiddie Schedule of Affective Disorders Scale (KSADS) used to evaluate for current and past depressive episode at each time point (interval between time points). Occurrence of first depressive episode was determined by the Depression Symptom Rating (DSR). We considered a score indicating at least sub-threshold major depression (a DSR of ≥3+) to be a depressive episode. DSR 4 and above and 5 alone will also be assessed.

SECONDARY OUTCOMES:
Depressed mood | 0, 2, 6, 12, 24 months
  The Center for Epidemiological Studies of Depression(CES-D)Scale -Change in CES-D score between groups (CATCH-IT & HEALTHED) across the duration of the study and for each assessment point
Vulnerability Factors | 0, 2, 6, 12, 18, 24 months
  Sibling Inventory of Differential Experience, (SIDE), Child/Parent Report of Parental Behavior Inventory (CRPBI - teen and parent), Conflict Behavior Questionnaire (CBQ - teen and parent), Beck Hopelessness Scale, Adolescent Life Events Questionnaire (ALEQ) (not all measures at all time points)
Quality of Life, educational impairment and other mental disorder symptoms or episodes | 0, 2, 6, 12, 18, 24 months
  Masten's Status Questionnaire,World Health Organization (WHO) Quality of Life Scale , Educational Impairment Scale, Change in scales of SCARED, Disruptive Behavior Disorder Scale (DBD - teen and parent), CRAFFT (substance abuse), SCARED (anxiety), Global Assessment Scale (GAS, assessor scores from KSADS responses) scores (not all measures at all time points).

OTHER OUTCOMES:
Adherence to Internet Use | continous measure
  Counting the number of logs/subject (over 2 years), number of characters typed, number of clicks in each page, time spent on each session and total time spent online and Socio-cultural Relevance Scale.
Implementation | 0, 2, 24 months
  Changes in perceived feasibility and implementation of the study from the healthcare professionals (physicians, nurse and leaders)from baseline to the completion of the study at 24 months.
Motivation (adolescent) | 0,2,12 months
  Theory of Planned Behavior Scale, Trans-Theoretical Model Scale
Demographic Information | 0,2,6,12,24 months
  assesses age, height, weight, contact information, race, ethnicity, home demographics, educational level of parents.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Van Voorhees, MD, MPH, Principal Investigator — UIC; Tracy Gladstone, PHD, Principal Investigator — Wellesley Center for Women
Locations (7):
- United States (7):
  - ACCESS Healthcare Systems, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Northshore Healthcare Systems, Evanston, Illinois
  - Advocate Health Care, Oak Lawn, Illinois
  - Children's Clinic, Oak Park, Illinois
  - Franciscan St. Margaret Health, Dyer, Indiana
  - Wellesley Center for Women, Wellesley, Massachusetts

REFERENCES:
- [Derived] Van Voorhees B, Gladstone TRG, Sobowale K, Brown CH, Aaby DA, Terrizzi DA, Canel J, Ching E, Berry AD, Cantorna J, Eder M, Beardslee W, Fitzgibbon M, Marko-Holguin M, Schiffer L, Lee M, de Forest SA, Sykes EE, Suor JH, Crawford TJ, Burkhouse KL, Goodwin BC, Bell C. 24-Month Outcomes of Primary Care Web-Based Depression Prevention Intervention in Adolescents: Randomized Clinical Trial. J Med Internet Res. 2020 Oct 28;22(10):e16802. doi: 10.2196/16802. PMID 33112254
- [Derived] Gladstone T, Buchholz KR, Fitzgibbon M, Schiffer L, Lee M, Voorhees BWV. Randomized Clinical Trial of an Internet-Based Adolescent Depression Prevention Intervention in Primary Care: Internalizing Symptom Outcomes. Int J Environ Res Public Health. 2020 Oct 22;17(21):7736. doi: 10.3390/ijerph17217736. PMID 33105889
- [Derived] Gladstone TG, Marko-Holguin M, Rothberg P, Nidetz J, Diehl A, DeFrino DT, Harris M, Ching E, Eder M, Canel J, Bell C, Beardslee WR, Brown CH, Griffiths K, Van Voorhees BW. An internet-based adolescent depression preventive intervention: study protocol for a randomized control trial. Trials. 2015 May 1;16:203. doi: 10.1186/s13063-015-0705-2. PMID 25927539